CLINICAL TRIAL: NCT01259648
Title: Randomized Study Evaluating the Efficacy and Safety of Remifentanil in a Rapid Sequence Induction for Fragile Subjects
Brief Title: Study Evaluating the Efficacy and Safety of Remifentanil in a Rapid Sequence Induction for Fragile Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LOCAL/2009/AC-02; 2009-018169-12 (EudraCT Number)
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2022-03

CONDITIONS: Tachycardia
Keywords: remifentanil; anesthesia induction; reactional tachycardia
MeSH Terms: conditions — Tachycardia | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.5 µg / kg remifentanil (Experimental): Induction anesthesia includes 0.5 µg/kg remifentanil in addition to classic induction anesthesia protocol.
  Interventions: Drug: 0.5 µg/kg remifentanil
- 1.0 µg/kg remifentanil (Experimental): Induction anesthesia includes 1.0 µg/kg remifentanil in addition to the classic induction protocol.
  Interventions: Drug: 1.0 µg/kg remifentanil
- NaCl (Placebo Comparator): An equivalent volume (1 ml for 10 kg of weight) of isotonic 0.9% NaCl is injected in addition to the classic anesthesia induction protocol
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: 0.5 µg/kg remifentanil — 0.5 µg/kg remifentanil is used during induction in addition to the classic induction protocol
  Arms: 0.5 µg / kg remifentanil
Drug: 1.0 µg/kg remifentanil — 1.0 µg/kg remifentanil is added to the classic induction anesthesia protocol
  Arms: 1.0 µg/kg remifentanil
Drug: NaCl — an equivalent volume (1 ml for 10 kg of weight) of 0.9% isotonic NaCl is injected in addition to the classic anesthesia induction protocol
  Arms: NaCl

SUMMARY:
The primary objective is to determine whether, during a rapid sequence intubation by etomidate, and succinylcholine Sellick maneuver, the administration of remifentanil at 2 different dosages (0.5 and 1.0 microgram per kg body weight), reduces potentially dangerous reactional tachycardia.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring rapid sequence intubation for whatever reason. This includes the following: a full stomach, obesity, diabetic gastroparesis, gastroesophageal reflux
* Patient able to give informed consent, and sign the consent.

Exclusion Criteria:

* Contraindication for the use of any drugs used (regardless of the patient group): a history of serious side effects, allergic reaction
* Morbid obesity (Body Mass Index > 40)
* Emergency situation with unstable hemodynamics, and stabilization is impossible before induction
* Inclusion in another research project within the past 3 months
* The patient is not insured or beneficiary of a health insurance plan (for the French centers)
* Patient under guardianship of any kind
* Patient unable to give informed consent
* Refusal to sign the consent form

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-03-09 (Actual); Primary Completion 2014-05-20 (Actual); Study Completion 2014-05-20 (Actual)

PRIMARY OUTCOMES:
Cardiac frequency (beats per minute) | 15 minutes
  Patient cardiac frequency (beats per minute) at the time of induction

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Chaumeron, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard
  - Polyclinique Grand Sud, Nîmes, Gard

IPD SHARING:
Plan to Share IPD: Yes
Data available upon request.

REFERENCES:
- [Result] Chaumeron A, Castanie J, Fortier LP, Basset P, Bastide S, Alonso S, Lefrant JY, Cuvillon P. Efficacy and safety of remifentanil in a rapid sequence induction in elderly patients: A three-arm parallel, double blind, randomised controlled trial. Anaesth Crit Care Pain Med. 2020 Apr;39(2):215-220. doi: 10.1016/j.accpm.2019.09.010. Epub 2019 Oct 12. PMID 31614244